CLINICAL TRIAL: NCT00804297
Title: Comparison of Octreotide and Standard Therapy vs. Standard Therapy Alone for the Treatment of Hypoglycemia in Patients Taking Sulfonylureas or a Combination of Insulin and Sulfonylureas Presenting to the Emergency Department
Brief Title: Octreotide for the Treatment of Sulfonylurea-Associated Hypoglycemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: (H)N-2877
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Hypoglycemia; Diabetes Mellitus
Keywords: Hypoglycemia; Diabetes Mellitus; Octreotide
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus | interventions — Octreotide; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Octreotide (drug)

SUMMARY:
Background:

Hypoglycemia is a common presentation to the Emergency Department. Management has traditionally involved rapid administration of IV 50% dextrose and dextrose containing IV fluids in addition to oral carbohydrates. Hypoglycemic patients taking only insulin can often times be treated as outlined above and safely discharged to home after a period of short observation in the Emergency Department. This procedure is also followed in the pre-hospital care arena, where insulin-dependent hypoglycemic patients are often treated and released.

In addition to diet-control and insulin, patients with diabetes maintain outpatient euglycemia with a class of drugs called sulfonylurea agents. This are believed to stimulate insulin release from pancreatic beta cells via a complex mechanism culminating in calcium influx and release of stored insulin from secretory granules within the pancreas. Whereas insulin-dependent diabetic patients are usually discharged home after establishing normal blood glucose levels, hospital admission is generally recommended in hypoglycemic patients taking oral sulfonylureas due to the long duration of effect and delayed clearance of the drugs and their metabolites and subsequent high likelihood of recurrent hypoglycemic episodes.

Octreotide is a somatostatin analog that is known to suppress numerous hormones including insulin. Dextrose itself induces insulin secretion thus theoretically contributing to rebound hypoglycemia when used to treat hypoglycemia. Octreotide is thought to block the elevated insulin levels that are a result of both the sulfonlyureas and dextrose. Recent case reports and one prospective study in healthy volunteers have demonstrated the safety and efficacy of octreotide administration for the treatment of sulfonylurea induced hypoglycemia. Based largely on the results of these studies some experts in field of toxicology have argued that administration of octreotide be standard therapy for all patients with recurrent hypoglycemic episodes who are known to be taking sulfonylureas.

Purpose:

Measure the difference in serum glucose and the incidence of hypoglycemia between two groups of sulfonylurea-dependent patients; a control group that receives standard therapy and an experimental group that receives standard therapy plus octreotide.

DETAILED DESCRIPTION:
Methods:

All adult (>18 years old) non-pregnant patients presenting to the Emergency Department with hypoglycemia (serum glucose < 60 mg/dl) will be identified and screened for inclusion by the ED physicians and research staff. Hypoglycemic patients whose glucose-control medications involve only insulin will be excluded. All patients whose medications involve oral sulfonlyureas or a combination of insulin and sulfonylureas will be asked to participate in this study. Patients will be required to read and sign an informed consent outlining the objectives and risks/ benefits of the proposed protocol. In addition to reading the consent, details of the study will be explained verbally by a trained emergency medicine research assistant and patients will be given the opportunity to have all their questions answered.

Study patients will be randomized to one of two treatment arms.

1. Standard treatment and placebo One ampule (50 mL) of IV 50% dextrose, oral carbohydrates and placebo (1cc of 0.9 % Normal Saline subcutaneuously) or
2. Standard treatment plus 75 micrograms octreotide subcutaneously.

Enrolled patients will not receive additional maintenance IV glucose fluids unless they become hypoglycemic (serum glucose < 60 mg/dL), in which case they will receive bolus doses of IV 50% dextrose and re-evaluated. All enrolled patients will be admitted to the hospital and monitored for recurrent hypoglycemic episodes. Bedside glucose determinations will be collected hourly for 4 hours followed by repeated calculations every 2 hours. Data points to be collected will include the mean serum glucose, number of hypoglycemic episodes (<60mg/dl) and total quantity of dextrose required to maintain euglycemia.

In the likely event that the hypoglycemia was diagnosed in the pre-hospital setting and the patient received IV 50% dextrose prior to arrival to the Emergency Department, a rapid bedside glucose determination will be obtained and if <60 mg/dl a second bolus of IV 50% dextrose given and the patient screened and approached about participation. If the emergency department serum glucose is >60mg/dl the patient will be screened and approached about participation without a second bolus of IV 50% dextrose.

ELIGIBILITY:
Inclusion Criteria:

Hypoglycemia (serum glucose < 60mg/dl) and concurrent use of a sulfonylurea.

Exclusion Criteria:

Age <18. Pregnancy. Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-06; Study Completion 2007-01

PRIMARY OUTCOMES:
mean glucose level for the non-octreotide group is higher than the octreotide group

SECONDARY OUTCOMES:
number of hypoglicemic events

CONTACTS AND LOCATIONS:
Overall Officials: Charles J Fasano, DO, Principal Investigator — Albert Einstein Medical Center
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States